CLINICAL TRIAL: NCT04368416
Title: Prevalence of Anxiety/Depression, Sleep Disturbances and Alcohol Use Disorder in Elderly With Cognitive Complaints
Brief Title: Anxiety/Depression, Sleep and Alcohol in Elderly Anxiety/Depression, Sleep Disturbances and Alcohol Use Disorder in Elderly With Cognitive Complaints
Acronym: MEM-ASA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A02928-49
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-02

CONDITIONS: Anxiety State; Sleep Disturbance; Alcohol Abuse; Aging; Dementia
MeSH Terms: conditions — Anxiety Disorders; Parasomnias; Alcoholism; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of MEM-ASA is to investigate the prevalence of anxiety/depression, sleep disturbances and alcohol use disorder in elderly with cognitive complaints.

In memory clinics of Normandy (France), all patients aged over 50 year-old are systematically questioned about anxiety, depression, sleep quality and alcohol use disorder. They also perform a neuropsychological assessment. Questionnaires are given to the patient and his/her caregiver to be filled in at home.

Levels of anxiety/depression, sleep quality and alcohol consumption are related to neuropsychological performance, diagnosis and responses to the questionaires.

ELIGIBILITY:
Inclusion Criteria:

* To have cognitive complaints
* To have french as native language
* Not to be opposed to be included
* To be affiliated to the social security

Exclusion Criteria:

-To be under tutorship or curatorship

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of memory clinics in Normandy.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety and depression | At inclusion
  Responses to questions during anamnesis
Sleep quality | At inclusion
  Responses to questions during anamnesis
Alcohol use disorder | At inclusion
  Responses to questions during anamnesis

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BRANGER, MD, Principal Investigator — CHU CAEN
Locations (1):
- University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No